CLINICAL TRIAL: NCT07245732
Title: STeroid Options for RA Management (STORM-RA): Oral Versus Intramuscular Steroid Use to Control Rheumatoid Arthritis Flares: A Pragmatic Randomized Clinical Trial
Brief Title: Oral Versus Intramuscular Steroid Use to Control Rheumatoid Arthritis Flares
Acronym: STORM-RA
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTO Project ID: 4847
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-10

CONDITIONS: Rheumatoid Arthritis (RA)
Keywords: Pragmatic trial; Qualitative study; Study within a trial (SWAT); Steroids; Rheumatoid arthritis; Quality of life; Disease flare; Patient reported outcomes; Adverse effects
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Glucocorticoids

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral (Experimental): Oral steroid arm: Prednisone 15 mg/day for a week, reducing by 5 mg/day every 7 days until tapered off
  Interventions: Drug: Glucocorticoid (GC)
- Intramuscular (Experimental): Single dose 120 mg intramuscular methylprednisolone to the deltoid
  Interventions: Drug: Glucocorticoid (GC)

INTERVENTIONS:
Drug: Glucocorticoid (GC) — * PO GC arm: Prednisone 15 mg/day for a week, reducing by 5 mg/day every 7 days until tapered off
  * IM GC arm: Single dose 120 mg IM methylprednisolone to the deltoid

SUMMARY:
People living with rheumatoid arthritis (RA) often experience flares-periods where their symptoms suddenly get worse. These flares can cause significant pain, make it harder to move and do daily activities, and lower overall quality of life. Doctors often treat flares with medications called glucocorticoids (GCs), which reduce inflammation. These medications can be taken by mouth (oral/PO) or given as a single injection into the muscle (intramuscular/IM). However, it's not clear which option works better from the patient's point of view-especially when it comes to relief of symptoms, improvements in function, and satisfaction with treatment. Most research so far has focused on how well the drugs control the disease, rather than how they impact the patient's overall experience.

Research Questions:

1. Does a single GC injection work just as well as taking pills over a few weeks in improving symptoms reported by patients?
2. How do the two treatments compare in terms of symptom relief, ability to function, and patient satisfaction?
3. What do patients think and feel about using GCs to treat RA flares?

What the Investigators Think:

The investigators believe that a one-time GC injection is just as good as taking pills for a few weeks when it comes to managing RA flares. In fact, the injection might even be safer and preferred by patients.

What the Investigators are Doing:

The investigators will study 220 adults with RA who are currently having a flare (with at least 3 swollen and tender joints). These patients will be recruited from rheumatology clinics at the University of Toronto and must not have used GCs in the past month. They will be randomly assigned to receive either:

A single injection (Methylprednisolone 120 mg), or Oral pills (Prednisone starting at 15 mg daily and tapering down over 3 weeks).

The main thing the investigators will look at is how much better patients feel after 6 weeks, based on a questionnaire designed to measure RA flares. The investigators will also look at how well they function, how satisfied they are with the treatment, and whether they had any side effects.

In addition, 20 patients (10 from each group) will be interviewed to understand their experiences and opinions about flare treatment in more detail.

Why This Is Possible:

The investigators have already surveyed University of Toronto rheumatologists who support the idea and provided input on study design. The investigators have also partnered with experts in research methods, national arthritis organizations, and patient groups to make sure the study is relevant and meaningful. Ethics approval has been obtained.

Why It Matters:

RA flares can have a major impact on people's lives. While current treatments help control inflammation, the investigators need to better understand how these treatments affect people from their own perspective. This study will shift the focus to what matters most to patients, helping doctors and patients choose the best treatment based not only on medical results but also on the patient's experience. This could lead to more effective and personalized care for people living with RA.

DETAILED DESCRIPTION:
Background Rheumatoid arthritis (RA) is a chronic inflammatory disorder that can severely impact patients' quality of life, with acute flares being a major challenge (1). These flares lead to pain, swelling, and functional limitations, affecting both physical and emotional well-being, and often result in treatment escalation and long-term complications (2,3). Despite their frequency, there is a gap in understanding optimal management strategies, particularly regarding glucocorticoid (GC) therapy.

Current guidelines recommend oral glucocorticoids (PO GC) as the standard treatment, typically as a tapering regimen, but intra-muscular (IM) injections are also used in practice (4,5). However, there is no direct comparison of their short-term effectiveness, safety, and patient experience. Without this evidence, clinicians lack guidance on which method best suits individual patients, especially regarding flare severity and disease activity.

Understanding the patient experience during RA flares is critical in guiding clinical decision-making. While disease activity measurements, such as the Disease Activity Score (DAS28), are commonly used to assess treatment response, they do not capture the full spectrum of the patient's lived experience during a flare. Patient-reported outcomes (PROs), including pain, fatigue, and overall well-being, are integral to understanding how patients perceive their condition and treatment efficacy (6). Incorporating PROs into clinical trials and practice will not only provide a more holistic view of treatment response but will also help to align these subjective experiences with traditional objective measures of disease activity (7). As such, evaluating the impact of different GC treatments on PROs is essential to determining the most effective approach for managing RA flares and improving patient outcomes.

This study aims to address this gap by conducting a comparative study of IM versus PO steroids for acute RA flare management, with a focus on patient reported outcomes (PROs). By incorporating PROs alongside traditional disease activity assessments, this study will provide a comprehensive understanding of how different treatment strategies impact both clinical and patient-centered outcomes. This patient-focused approach has the potential to significantly influence treatment guidelines and improve the overall management of RA flares.

Aim: To compare the effectiveness of IM versus PO GC in improving patient-reported symptoms of RA flares.

Objectives: In patients with established RA experiencing a flare, the investigators aim:

1. To assess whether IM GC administration is non-inferior to PO GC administration in improving RA flare symptoms.
2. To evaluate differences between IM and PO GC in terms of clinical efficacy, functional improvements, treatment satisfaction and side effects in RA patients experiencing flares.
3. To qualitatively analyze the attitudes, preferences and treatment priorities regarding IM versus PO GC use for RA flares

Hypotheses: The investigators hypothesize that a single IM GC dose will be non-inferior to a PO regimen for improving acute RA flare symptoms, as measured by the RA-FQ score. While the investigators do not expect major differences in disease activity score improvements between arms, the investigators anticipate that IM administration may offer advantages through a lower cumulative steroid exposure, potentially improving the safety profile. In addition, the investigators expect higher patient satisfaction and preference with the IM approach, given the convenience of a one-time, physician-administered treatment compared to a 21-day daily PO regimen.

Research Approach/Methodology and Rationale

Project Design This will be a 3-year, prospective, pragmatic, non-inferiority, randomized controlled trial (RCT). Unlike traditional explanatory RCTs, which evaluate interventions under ideal conditions, the proposed study's pragmatic design reflects real-world practice to enhance the external validity of the results (8). Additionally, a Study Within a Trial (SWAT) will be conducted, involving a subgroup of 20 patients (10 per arm) who will participate in semi-structured interviews to explore patient perspectives on managing RA flares. This non-inferiority study design is predicated on the investigators' hypothesis that a single IM GC dose is non-inferior to PO GC for RA flare symptom improvement.

Study population Adult patients ≥18 years of age, who fulfill ACR/EULAR 2010 classification criteria with an established diagnosis of RA and experiencing a flare will be recruited from five rheumatology clinics at the University of Toronto (9). The investigators will include consecutive patients who have symptoms of an RA flare defined as ≥3 swollen and ≥3 tender joints, for which the treating rheumatologist would have otherwise prescribed systemic GC.

Study Interventions

The following interventions are proposed to be randomized in a 1:1 fashion:

* PO GC arm: Prednisone 15 mg/day for a week, reducing by 5 mg/day every 7 days until tapered fully off
* IM GC arm: Single dose 120 mg IM methylprednisolone

Given the pragmatic nature of this study, treating rheumatologists will have the flexibility to adjust, switch, or modify the doses of any DMARD therapy or non-steroidal anti-inflammatory drugs (NSAIDs) as part of routine care at any point after the intervention is administered.

Randomization The calculated sample size will be 101 patients per group. Assuming approximately 10% attrition, the investigators aim to recruit 220 patients. The investigators will use block randomization within the 5 sites with random block sizes to minimize selection bias (10).

Primary Outcome Measure The primary outcome measure will focus on the impact of GC therapy on the RA flare experience. The investigators will use the Rheumatoid Arthritis Flare Questionnaire (RA-FQ), a 5-item questionnaire developed by the OMERACT RA Flare Group in 2016, to assess pain, fatigue and functional limitations during a flare. The RA-FQ has been validated for content, face validity, construct validity shows sensitivity to change (11,12).

Secondary Outcome Measures. The investigators will explore additional outcomes that are standard endpoints in RA trials. These will provide insights into clinical efficacy, safety, and patient experiences with GC treatments.

1. Clinical Disease Activity Index (CDAI) difference at 6 weeks: This will assess RA disease activity to provide a clinical response anchor, as the RA-FQ has not been extensively studied in GC trials for RA.
2. Glucocorticoid adverse effects: Data on adverse events (AEs) will be collected via physician report at week 6.
3. Systemic GC use between 6 and 12 weeks: The investigators will assess whether the IM and PO routes of GC administration offer advantages in minimizing GC use beyond the 6-week trial period.
4. Treatment Satisfaction Questionnaire for Medication (TSQM) difference at 6 weeks: The TSQM v1.4, a PRO used in prior RA studies, will measure patient satisfaction with the treatment (13).
5. Health Assessment Questionnaire Disability Index (HAQ-DI): The HAQ-DI will capture functional changes between therapies, given its robust psychometric properties and responsiveness to disease activity (14).
6. Qualitative study outcome: A qualitative component will explore patient perspectives on IM versus PO GC for flare management. Using qualitative description, the investigators will identify common themes across participants to inform clinical practice (15). The investigators aim to recruit 20 participants (10 per group) to achieve conceptual thematic saturation.

Analytic Plan

Sample size The investigators calculated the sample size for the primary outcome based on non-inferiority in RA-FQ score changes at 6 weeks between the IM and PO groups. Using CATCH data showing a RA-FQ improvement of 10.0±14.2 (unpublished), the investigators set a non-inferiority margin of -5.0, per FDA guidelines (16). With 80% power and alpha of 0.05, 101 patients per group are needed. Factoring in 10% attrition, the investigators aim to recruit 220 patients.

Statistical Analyses Patient demographic and clinical characteristics will be summarized and compared by randomization groups, including age, sex, race, RF/CCP positivity, disease and flare duration, prior DMARD/NSAID use, co-morbidities, erosions, and CRP. For the primary outcome (RA-FQ scores), an ANCOVA linear model will adjust for baseline RA-FQ scores, NSAID and DMARD use, and study site (17). Given the pragmatic trial design, NSAID and DMARD use will be allowed, and adjusted for as potential confounders. Intention-to-treat analysis will be used, with per-protocol analysis as a sensitivity analysis. Secondary outcomes (CDAI, TSQM, additional GCs by 12 weeks, HAQ-DI, and adverse effects) will be compared descriptively. The qualitative component will use descriptive analysis to capture patients' experiences with RA flare treatments (IM vs. PO GC), maintaining minimal interpretation and grounded in an inductive, interpretivist approach (15). This will provide insights into patient preferences for flare management.

Potential to create new knowledge The patient experience is at the epicenter of RA flare management and treatment evaluation. Therefore, the focus of this proposed research project will be aimed towards the patient's flare experience, incorporating the use of PROs in both its primary and secondary outcomes, as well as additionally employing a qualitative study within a trial design to illuminate patient viewpoints on the preferences of people living with RA around treatment of flares, with a focus on use of steroids. Evaluating the comparative effectiveness of various GC formulations and dosages will help address the knowledge gaps in current clinical practice on the preferred route and dosage of GCs to optimize safety and effectiveness.

Furthermore, the significance of this study extends beyond its direct outcomes. It will assess the feasibility of conducting a pragmatic clinical trial within an academic network, combining insights from clinicians, researchers and patient partners. The investigators hope that lessons learned from this study can be applied to answer other clinically relevant rheumatology questions in the real-world setting. Given many trials exclude patients with comorbidities or are restricted to testing novel therapies, this framework provides an opportunity to test "real problems" affecting "real patients."

Given the global prevalence of RA and associated flares, alongside the ongoing debate over the optimal route of GC administration, the study's findings hold considerable international relevance. This study has the potential to reshape paradigms in flare management, potentially revolutionizing future approaches to RA treatment worldwide.

ELIGIBILITY:
Inclusion Criteria:

* Rheumatologist verified RA diagnosis.
* Patients are allowed to be on non-steroidal anti-inflammatory drugs (NSAIDs) prior to randomization, but the dosages must be stable for ≥2 weeks prior to randomization.
* Patients must be on stable doses of conventional synthetic disease-modifying antirheumatic drugs (csDMARD)/targeted synthetic disease-modifying antirheumatic drugs (tsDMARD)/biologics (bDMARDs) for ≥8 weeks prior to randomization.

Exclusion Criteria:

* Allergies, intolerances or contraindications to systemic GCs or IM injections
* Patients with active malignancy, are pregnant or breastfeeding.
* Patients who have received systemic or intra-articular GC within 4-weeks of randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2029-03 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
Rheumatoid Arthritis Flare Questionnaire (RA-FQ) | Weeks 0, 1, 2, 4, 6 (primary outcome at 6-weeks)
  The Rheumatoid Arthritis Flare Questionnaire (RA-FQ) was created and endorsed in 2016 by OMERACT to assess flare treatment response over time, addressing many of the shortcomings associated with the use of disease activity measure scores to gauge flare evolution. The RA-FQ includes five patient-reported items-pain, physical function, stiffness, fatigue, and participation-rated on an 11-point scale over the past week, producing a total score from 0 to 50, with higher scores indicating worse flare disease activity. Validated for content and construct validity, the RA-FQ is sensitive to change within one week and aligns well with the Clinical Disease Activity Index (CDAI), making it a practical, patient-centered tool with strong clinical relevance.

SECONDARY OUTCOMES:
Health Assessment Questionnaire Disability Index (HAQ-DI) | Weeks 0 and 6
  The HAQ-DI, a widely used self-report tool in RA, assesses functional ability in daily activities on a 0-3 scale (higher scores indicate greater disability). Given its ease of use and strong psychometric properties, it was chosen to detect therapy-related changes, as it is sensitive to disease activity fluctuations.
Clinical Disease Activity Index (CDAI) | Weeks 0 and 6
  The investigators selected the CDAI to anchor clinical response, as the RA-FQ is not well studied in GC trials. The CDAI, which is endorsed by the American College of Rheumatology, combines joint counts with patient and physician global assessments and is practical for clinical use, requiring no laboratory tests-an advantage in the pragmatic trial design. The scores range from 0 to 76, with high scores indicating higher disease activity.
Glucocorticoid adverse events | 6-weeks
  The investigators will collect data at each in-person clinical visit on adverse events (AEs). Serious AEs will be defined according to the Medical Dictionary for Regulatory Activities (MedDRA).
Systemic GC use between 6 and 12 weeks | 6 to 12-weeks
  We will assess whether IM or PO GC administration reduces GC use beyond the 6-week trial by collecting data at 12 weeks post-randomization on additional GC requirements.
Treatment Satisfaction Questionnaire for Medication (TSQM) | Weeks 0 and 6
  The TSQM v1.4 is a validated PRO measuring treatment satisfaction in chronic diseases, including RA. It covers Effectiveness, Side Effects, Convenience, and Global Satisfaction, with scores from 0 to 100 where scores ≥80 indicate good satisfaction.

CONTACTS AND LOCATIONS:
Locations (5):
- Canada (5):
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Women's College Hospital, Toronto, Ontario
  - Toronto Western Hospital, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wang B, Ogburn EL, Rosenblum M. Analysis of covariance in randomized trials: More precision and valid confidence intervals, without model assumptions. Biometrics. 2019 Dec;75(4):1391-1400. doi: 10.1111/biom.13062. Epub 2019 Jun 3. PMID 31009064
- [Background] King LK, Mahmoudian A, Waugh EJ, Stanaitis I, Gomes M, Hung V, MacKay C, Liew JW, Wang Q, Turkiewicz A, Haugen IK, Appleton CT, Lohmander S, Englund M, Runhaar J, Neogi T, Hawker GA; OARSI Early-stage Symptomatic Knee Osteoarthritis Initiative. "You don't put it down to arthritis": A qualitative study of the first symptoms recalled by individuals with knee osteoarthritis. Osteoarthr Cartil Open. 2023 Dec 16;6(1):100428. doi: 10.1016/j.ocarto.2023.100428. eCollection 2024 Mar. PMID 38229918
- [Background] Looijen AEM, van Mulligen E, Vonkeman HE, van der Helm-van Mil AHM, de Jong PHP. Responsiveness and sensitivity of PROMs to change in disease activity status in early and established rheumatoid arthritis. Rheumatology (Oxford). 2025 Mar 1;64(3):1060-1067. doi: 10.1093/rheumatology/keae213. PMID 38574380
- [Background] Radawski C, Genovese MC, Hauber B, Nowell WB, Hollis K, Gaich CL, DeLozier AM, Gavigan K, Reynolds M, Cardoso A, Curtis JR. Patient Perceptions of Unmet Medical Need in Rheumatoid Arthritis: A Cross-Sectional Survey in the USA. Rheumatol Ther. 2019 Sep;6(3):461-471. doi: 10.1007/s40744-019-00168-5. Epub 2019 Aug 6. PMID 31385264
- [Background] Bartlett SJ, Bykerk VP, Schieir O, Valois MF, Pope JE, Boire G, Hitchon C, Hazlewood G, Bessette L, Keystone E, Thorne C, Tin D, Bingham CO 3rd; CATCH Investigators. "From Where I Stand": using multiple anchors yields different benchmarks for meaningful improvement and worsening in the rheumatoid arthritis flare questionnaire (RA-FQ). Qual Life Res. 2023 May;32(5):1307-1318. doi: 10.1007/s11136-022-03227-7. Epub 2022 Sep 8. PMID 36074252
- [Background] Bartlett SJ, Barbic SP, Bykerk VP, Choy EH, Alten R, Christensen R, den Broeder A, Fautrel B, Furst DE, Guillemin F, Hewlett S, Leong AL, Lyddiatt A, March L, Montie P, Pohl C, Scholte Voshaar M, Woodworth TG, Bingham CO 3rd. Content and Construct Validity, Reliability, and Responsiveness of the Rheumatoid Arthritis Flare Questionnaire: OMERACT 2016 Workshop Report. J Rheumatol. 2017 Oct;44(10):1536-1543. doi: 10.3899/jrheum.161145. Epub 2017 Aug 15. PMID 28811351
- [Background] Efird J. Blocked randomization with randomly selected block sizes. Int J Environ Res Public Health. 2011 Jan;8(1):15-20. doi: 10.3390/ijerph8010015. Epub 2010 Dec 23. PMID 21318011
- [Background] Aletaha D, Neogi T, Silman AJ, Funovits J, Felson DT, Bingham CO 3rd, Birnbaum NS, Burmester GR, Bykerk VP, Cohen MD, Combe B, Costenbader KH, Dougados M, Emery P, Ferraccioli G, Hazes JM, Hobbs K, Huizinga TW, Kavanaugh A, Kay J, Kvien TK, Laing T, Mease P, Menard HA, Moreland LW, Naden RL, Pincus T, Smolen JS, Stanislawska-Biernat E, Symmons D, Tak PP, Upchurch KS, Vencovsky J, Wolfe F, Hawker G. 2010 rheumatoid arthritis classification criteria: an American College of Rheumatology/European League Against Rheumatism collaborative initiative. Ann Rheum Dis. 2010 Sep;69(9):1580-8. doi: 10.1136/ard.2010.138461. PMID 20699241
- [Background] Ford I, Norrie J. Pragmatic Trials. N Engl J Med. 2016 Aug 4;375(5):454-63. doi: 10.1056/NEJMra1510059. No abstract available. PMID 27518663
- [Background] Kluzek S, Dean B, Wartolowska KA. Patient-reported outcome measures (PROMs) as proof of treatment efficacy. BMJ Evid Based Med. 2022 Jun;27(3):153-155. doi: 10.1136/bmjebm-2020-111573. Epub 2021 Jun 4. No abstract available. PMID 34088713
- [Background] Orbai AM, Bingham CO 3rd. Patient reported outcomes in rheumatoid arthritis clinical trials. Curr Rheumatol Rep. 2015 Apr;17(4):28. doi: 10.1007/s11926-015-0501-8. PMID 25854489
- [Background] Nikolic RPA, Pardo JP, Pope JE, Barber CEH, Barnabe C, Schieir O, Jamal S, Legge A, Kuriya B, Akhavan P, Thorne JC, Bombardier C, Taylor-Gjevre R, Bykerk V, Khraishi M, Proulx L, Richards DP, Tugwell P, Agarwal A, Bansback N, Hazlewood GS. Canadian Rheumatology Association Living Guidelines for Rheumatoid Arthritis: Update #2. J Rheumatol. 2024 Sep 1;51(9):940-941. doi: 10.3899/jrheum.2024-0540. No abstract available. PMID 39009382
- [Background] Smolen JS, Landewe RBM, Bergstra SA, Kerschbaumer A, Sepriano A, Aletaha D, Caporali R, Edwards CJ, Hyrich KL, Pope JE, de Souza S, Stamm TA, Takeuchi T, Verschueren P, Winthrop KL, Balsa A, Bathon JM, Buch MH, Burmester GR, Buttgereit F, Cardiel MH, Chatzidionysiou K, Codreanu C, Cutolo M, den Broeder AA, El Aoufy K, Finckh A, Fonseca JE, Gottenberg JE, Haavardsholm EA, Iagnocco A, Lauper K, Li Z, McInnes IB, Mysler EF, Nash P, Poor G, Ristic GG, Rivellese F, Rubbert-Roth A, Schulze-Koops H, Stoilov N, Strangfeld A, van der Helm-van Mil A, van Duuren E, Vliet Vlieland TPM, Westhovens R, van der Heijde D. EULAR recommendations for the management of rheumatoid arthritis with synthetic and biological disease-modifying antirheumatic drugs: 2022 update. Ann Rheum Dis. 2023 Jan;82(1):3-18. doi: 10.1136/ard-2022-223356. Epub 2022 Nov 10. PMID 36357155
- [Background] Alten R, Pohl C, Choy EH, Christensen R, Furst DE, Hewlett SE, Leong A, May JE, Sanderson TC, Strand V, Woodworth TG, Bingham CO 3rd; OMERACT RA Flare Definition Working Group. Developing a construct to evaluate flares in rheumatoid arthritis: a conceptual report of the OMERACT RA Flare Definition Working Group. J Rheumatol. 2011 Aug;38(8):1745-50. doi: 10.3899/jrheum.110400. PMID 21807796
- [Background] Flurey CA, Morris M, Richards P, Hughes R, Hewlett S. It's like a juggling act: rheumatoid arthritis patient perspectives on daily life and flare while on current treatment regimes. Rheumatology (Oxford). 2014 Apr;53(4):696-703. doi: 10.1093/rheumatology/ket416. Epub 2013 Dec 19. PMID 24357813
- [Background] Smolen JS, Aletaha D, Barton A, Burmester GR, Emery P, Firestein GS, Kavanaugh A, McInnes IB, Solomon DH, Strand V, Yamamoto K. Rheumatoid arthritis. Nat Rev Dis Primers. 2018 Feb 8;4:18001. doi: 10.1038/nrdp.2018.1. PMID 29417936

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-03-24): https://cdn.clinicaltrials.gov/large-docs/32/NCT07245732/Prot_SAP_000.pdf
  • Informed Consent Form (2025-10-08): https://cdn.clinicaltrials.gov/large-docs/32/NCT07245732/ICF_001.pdf